CLINICAL TRIAL: NCT07023497
Title: Determination of the Optimal Dose of Intrathecal Morphine for Postoperative Analgesia After Cesarean Section Using the Up-and-Down Sequential Allocation Method
Brief Title: Determining the Optimal Dose of Intrathecal Morphine for Post-Cesarean Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Agathi Karakosta, Assistant Professor of Anaesthesiology, University of Ioannina
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8-1-2024/489
Record Dates: First submitted 2025-06-07; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Morphine; Cesarean Section; Postoperative Pain, Acute; Spinal Analgesia; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: We aim to employ an up-and-down sequential allocation method, a prospective, non-randomized, double-blind design commonly used in dose-finding studies. Each participant receives a dose of intrathecal morphine based on the analgesic response of the previous participant: the dose is increased following inadequate analgesia and decreased following effective pain relief.
Masking Description: This is a single-arm dose-finding study using a double-blind design. The participant and outcome assessor are blinded to the morphine dose administered, but all participants receive the same intervention (intrathecal morphine) with dose variation based on sequential allocation. No multi-arm comparison is involved.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-Finding Arm (Experimental): Participants receive spinal anesthesia with a fixed dose of fentanyl and ropivacaine, and a variable dose of morphine determined by the up-and-down sequential allocation method.
  Interventions: Drug: Intrathecal morphine

INTERVENTIONS:
Drug: Intrathecal morphine — Intrathecal morphine with fixed-dose fentanyl and ropivacaine

SUMMARY:
Using spinal or epidural anesthesia (known as neuraxial blocks) is the gold standard for pain control during childbirth, especially in cesarean sections (C-sections). However, many women experience moderate to severe pain after a C-section, which can affect both their physical and emotional well-being, and even impact their ability to care for their newborn. Unfortunately, this pain is often not treated effectively, which can lead to increased sensitivity to pain or even chronic postoperative pain.

One effective way to manage this pain is by giving opioids directly into the spinal fluid (subarachnoid space). This method allows doctors to use much smaller doses than would be needed if the same medication were given through a vein, which also helps avoid many of the common side effects of opioids like respiratory depression, nausea, pruritus, and constipation.

Common opioids used in this setting include fentanyl, sufentanil, and morphine. These drugs behave differently depending on their chemical properties. For example, drugs that are more fat-soluble work faster, while those that are less fat-soluble tend to last longer. Morphine, which is less fat-soluble than the others, provides strong and long-lasting pain relief. When injected spinally, its effect can last 18-24 hours, with the pain relief starting 1-2 hours after the injection. Its performance is comparable to that of epidural anesthesia or nerve blocks.

Researchers have studied a wide range of spinal morphine doses (from 20 to 500 micrograms) to find the most effective and safest dose. Most of these studies are small or use set doses without clear reasoning. Recently, a method called sequential allocation has become popular for finding the best dose more accurately.

About the Study This research aims to find the ideal dose of spinal morphine when it's given with a fixed amount of fentanyl and varying doses of ropivacaine (a local anesthetic) during spinal anesthesia for C-section in healthy full-term parturients. The goal is to find the dose that provides adequate analgesia (pain score under 3 out of 10) for at least 12 hours after surgery.

This is a prospective, non-randomized, double-blind study. The study follows ethical standards and all participants sign an informed consent form. Two anesthesiologists are involved in each case: one handles the spinal injection and dose decision (based on the previous patient's response), while the other monitors the patient and collects the data without knowing the dose used.

Anesthetic Technique Spinal anesthesia is done using standard procedures. A very fine needle (25 or 27 gauge) is used to inject a mixture of fentanyl (15 mcg), a variable dose of ropivacaine (based on somatometrics), and a variable dose of morphine (based on the algorithm). The mixture is injected slowly (1 ml every 10 seconds), with the needle facing toward the head. After surgery, all women receive additional pain medications like paracetamol and NSAIDs as part of a multimodal pain relief approach.

How the Morphine Dose is Decided

The dose of morphine changes based on whether the previous participant had effective pain relief. Pain relief is considered successful if the pain score stays at or below 3 (on a 0-10 scale) for at least 12 hours after the spinal injection. For the first woman in the study, the starting dose is chosen based on published research. Then:

* If the previous participant had good pain control (NRS ≤3 for 12 hours), the dose for the next woman is reduced by 20 micrograms.
* If pain control was poor (NRS >3 within the first 12 hours), the dose is increased by 40 micrograms.

This up-and-down adjustment continues for each new participant.

DETAILED DESCRIPTION:
Introduction Neuraxial blocks, including epidural or spinal anesthesia/analgesia are the gold standard in obstetric anesthesia. Particularly, regional anesthesia is recommended for parturients undergoing elective cesarean sections (C-sections) because it is safer and leads to reduced maternal and neonatal morbidity compared to general anesthesia. C-sections are associated with moderate to severe postoperative pain in a significant percentage of women, which can have physical and psychological effects on both the mother and the newborn. Postoperative pain following a C-section is often undertreated, potentially leading to hyperalgesia, persistent acute pain, or even chronic postoperative pain. The administration of opioids via the subarachnoid route is an important tool for anesthesiologists in managing acute postoperative pain after C-sections, providing satisfactory analgesic effects. This method allows for a significant reduction in the dosage required compared to intravenous administration needed to achieve the same analgesic effect, thereby avoiding the side effects associated with opioids, such as respiratory depression, opioid-induced hyperalgesia, postoperative nausea/vomiting, pruritus, bowel obstruction, and others. Fentanyl, sufentanil, and morphine are common opioids frequently used in obstetric anesthesia/analgesia. The action of these substances depends on their physicochemical properties. The greater the lipophilicity of an opioid, the faster its onset of action, and the smaller its partition coefficient, the longer its duration of action. Morphine is the drug that exhibits the strongest and most prolonged effect, as it has the lowest lipophilicity among the commonly administered opioids. After administration, its concentration in the CSF remains stable with a gradual decrease after the first twelve hours. The onset of action following subarachnoid administration is estimated to be 1-2 hours, and its analgesic effect, which is clearly superior compared to other routes of administration (intravenous, intramuscular, or subcutaneous), is reported to be comparable to that of epidural anesthesia (EA) and paravertebral blocks, lasting from 18 to 24 hours.

The optimal dose of morphine for intrathecal administration remains a popular topic in published literature, with numerous studies examining a dose range from 25 to 500 µg. Most of these studies are observational or comparative, with limitations such as the use of arbitrarily defined doses and small sample sizes.

The sequential allocation methodology for assessing the dose-response relationship is gaining popularity in anesthesiology overall, including in obstetric anesthesia. Specifically, only few studies have incorporated this methodology, each with its own limitations, such as small sample sizes and differing study designs (i.e., comparing different opioids or evaluating analgesic efficacy only in vaginal delivery and not in cesarean section).

Aim of the study The current research protocol aims to investigate the dose-response relationship for morphine when co-administered with a fixed dose of fentanyl and a variable dose of ropivacaine in healthy term parturients scheduled for cesarean section. This approach may provide valuable data for a better understanding of the analgesic effects of morphine in clinical practice.

Study Objective The primary objective of this study is to determine the dose-response relationship of intrathecally administered morphine in healthy term parturients scheduled to undergo cesarean section under single-shot spinal anesthesia. The effective dose of morphine is defined as the dose that provides satisfactory analgesia (Numerical Rating Scale <3/10) at least 12 hours after intrathecal administration. The dose-response relationship of morphine will be described by determining the ED50 and ED90 (median effective dose and 90% effective dose). Secondary objectives of the study include assessing the time until rescue analgesia is administered, the total analgesic consumption during the first 24 hours postoperatively, the duration of sensory and motor blockade, the Apgar score of the newborn, intraoperative complications (such as discomfort, nausea, vomiting, and pruritus), maternal satisfaction, and postoperative complications related to anesthesia (such as pruritus, nausea/vomiting, ileus, sedation, headache, etc.).

Materials and Methods This study is a prospective, non-randomized, double-blind trial involving healthy parturients at term who are scheduled to undergo cesarean section under spinal anesthesia. The study will be conducted in full agreement with the principles of the Helsinki Declaration for clinical research, and candidates will be fully informed about the research protocol. Participants will sign a specific "informed consent" form. According to the protocol, two anesthesiologists are required to conduct the study: the principal investigator, who determines the morphine dose for each case based on the sequential allocation algorithm and performs the spinal anesthesia, and a second anesthesiologist, responsible solely for documenting postoperative study parameters and remaining blinded to the administered dose.

Anesthetic Technique The preoperative and intraoperative management of participants will follow the standard protocols of the clinic. The regional anesthesia technique to be applied is spinal anesthesia. With the parturient in a seated position, the O2-O3 or O3-O4 intervertebral space is identified. After skin antisepsis and local infiltration with lidocaine, a spinal injection of a mixture of local anesthetics and opioids will be performed. A pencil point needle, either 25 or 27 gauge, will be used for locating the subarachnoid space and injecting the anesthetic mixture. The administered anesthetic mixture will include a fixed dose of fentanyl (15 μg), a variable dose of ropivacaine based on the parturient's somatometric characteristics, and a variable dose of morphine according to the sequential allocation algorithm. The injection of the anesthetic mixture will be performed at a rate of approximately 1 ml of solution every 10 seconds, with the needle orifice directed cephalad.

Determination of Morphine Dose - Sequential Allocation Algorithm The morphine dose for each case is determined based on the response of the previous parturient to a higher or lower dose, following the sequential allocation algorithm. An exception is made for the first parturient participant in the study, for whom the initial morphine dose will be 100μg, based on literature data. For each subsequent case (excluding the first), the morphine dose will be adjusted, depending on the outcome of the postoperative analgesia of the previous participant. This outcome is classified as either "success" or "failure," whereby the morphine dose for the next participant will be decreased by 20 μg or increased by 40 μg, respectively.

Definition of Successful Postoperative Analgesia

Successful postoperative analgesia is defined as a numerical rating scale (NRS) of less than or equal to 3 (NRS≤3) for at least 12 hours following the spinal injection. According to the above definition, there are three possible scenarios:

1. Successful postoperative analgesia. NRS≤3 for at least 12 hours following the spinal injection. In this case, the dose of morphine for the next participant is reduced by 20 μg.
2. Unsuccessful postoperative analgesia. NRS>3 at any point during the first 12 hours following the spinal injection. In this case, the dose of spinal morphine for the next participant is increased by 40 μg.
3. Exclusion from the Study. Any deviation from the initial anesthesia plan, such as complications requiring reoperation or systemic medical intervention to manage anesthesia-related adverse effects (e.g., respiratory depression), at any point from the time of spinal injection up to 24 hours later constitutes a reason for exclusion from the study. In such cases, the same dose of morphine will be repeated in the next participant.

For safety reasons, the maximum allowable limit of spinally administered morphine will not exceed 300 μg. If a participant receives 300 μg of spinal morphine and has "unsuccessful" postoperative analgesia, the same dose will be repeated in the next participant.

Data Collection In the preoperative assessment, the medical history of the mother will be recorded, including age, somatometric characteristics, ASA (American Society of Anesthesiologists, physical status classification), and current medication. The obstetric history will also be documented, covering the number of births, number of pregnancies, gestational age, and the reason for surgical delivery (diagnosis). Intraoperatively, data will be collected on the duration of the block, which will be evaluated using hot-cold sensation tests, pinprick tests, and recording of the modified Bromage scale at both the onset and regression of the block. Additionally, the duration of surgery and any intraoperative events (e.g., hemodynamic instability, adverse effects related to administered medications, etc.) will be documented, along with any supplementary medications (type and dosage). The intensity of acute postoperative pain will be recorded using the NRS scale, along with any potential adverse effects related to anesthesia (as mentioned above). Specifically, monitoring of the aforementioned variables of interest will occur at 2, 6, 12, 16, and 24 hours after the spinal injection. Furthermore, patient satisfaction will be recorded using a validated tool at the 24-hour mark, assessed by a healthcare provider not involved in the study.

Sample Size and Statistical Analysis To determine the effective dose, the up-and-down sequential allocation method described by Dixon and Massey was used. This approach is widely applied for estimating the median effective dose (ED₅₀), as it provides statistically reliable results with a relatively small sample size; typically, 20 to 40 participants. However, this method primarily gathers data around ED₅₀ and is insufficient for estimating higher efficacy levels such as ED₉₀. For accurate ED₉₀ estimation, a second series of participants will be enrolled, starting from the previously estimated ED₅₀, to collect data in the upper range of the dose-response curve. The required sample size for ED₉₀ estimation will be determined following the calculation of ED₅₀.

Data analysis will be conducted using Stata™ software (Version 10.1 MP, Stata Corporation, College Station, TX 77845, USA).

ELIGIBILITY:
Inclusion Criteria:

* term parturient
* single pregnancy
* elective cesarean delivery
* adult parturient
* ASA II

Exclusion Criteria:

* participants under the age of 18
* extreme somatometric characteristics
* lack of patient consent
* absolute contraindications for spinal anesthesia
* urgent cesarean section
* presence of known fetal anomalies
* onset of labor prior to administration of the block
* history of chronic pain
* use of opioids (systemic or otherwise) for any reason (e.g., chronic malignant pain)
* communication difficulties (e.g., language barriers, cognitive impairments)
* allergy or hypersensitivity to morphine
* severe arrhythmia or other serious cardiovascular conditions
* severe hepatic or renal insufficiency

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving adequate postoperative analgesia within 12 hours after spinal injection | 0 to 24 hours post spinal anesthesia
  Adequate analgesia is defined as a Numerical Rating Scale (NRS, 0 to 10) pain score ≤3, maintained for at least 12 hours following intrathecal morphine administration for cesarean section. Each participant's outcome (success or failure) guides the dose selection for the next participant in accordance with the up-and-down sequential allocation method. The primary objective is to determine the ED50 and ED90 (median and 90% effective dose) of intrathecal morphine.

SECONDARY OUTCOMES:
Total analgesic consumption | 0 to 24 hours post surgery
  Cumulative dose of all systemic analgesics (opioids and non-opioids) administered during the first 24 hours postoperatively, recorded in morphine milligram equivalents (MME) where applicable.
Duration of sensory block | Intraoperative to early postoperative period (up to 6 hours)
  Time interval from spinal injection to full regression of sensory block to S2 dermatome, assessed using pinprick or cold test.
Duration of motor block | Intraoperative to early postoperative period (up to 6 hours)
  Time from spinal injection to complete recovery of motor function (Bromage score 0).
Neonatal Apgar Score | 1 and 5 minutes post-delivery
  Apgar score assessed at 1 and 5 minutes after birth to evaluate newborn status.
Maternal satisfaction | At 24 hours postoperatively
  Maternal satisfaction with anesthesia and pain management, assessed using a structured three-question questionnaire based on a 5-point Likert scale each.
Postoperative pruritus | 0 to 24 hours post spinal anesthesia
  Incidence of postoperative nausea and vomiting, measured on a scale from 0 (no nausea) to 4 (continuous episodes of vomiting).
Postoperative ileus | 0 to 24 hours post spinal anesthesia
  Incidence of postoperative ileus, recorded as a binary variable (yes/no).
Postoperative sedation | 0 to 24 hours post spinal anesthesia
  Incidence of sedation, as defined by the Ramsay Sedation Scale, ranging from 1 (anxious, agitated, or restless) to 6 (no response to stimulus).
Post-dural puncture headache | 0 to 24 hours post spinal anesthesia
  Incidence of post-dural puncture headache, recorded as a binary variable (yes/no).
Postoperative respiratory depression | 0 to 24 hours post spinal anesthesia
  Incidence of postoperative respiratory depression, defined as a respiratory rate of fewer than 8 breaths per minute and/or oxygen desaturation (SpO₂ <94%), was recorded as a binary variable (yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Undecided